CLINICAL TRIAL: NCT02205268
Title: A Pilot Study of Near Infrared Spectroscopy Neurofeedback Training of Prefrontal Cortex in Attention Deficit Hyperactivity Disorder
Brief Title: Near Infrared Spectroscopy Neurofeedback Training for ADHD
Acronym: ADHDNTx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Essex Partnership NHS Foundation Trust (Other Government)
Collaborators: University College, London (Other); Hertfordshire Community NHS Trust (Unknown)
Responsible Party: Principal Investigator, Dr Thomas Dannhauser, Chief Investigator, North Essex Partnership NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEPADHDNTX
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit Disorder with Hyperactivity; Attention Deficit Hyperactivity Disorder; Biofeedback; Neurofeedback Training; Prefrontal Cortex; Near infrared spectroscopy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neurofeedback training (Experimental): 20 sessions of near infrared spectroscopy neurofeedback training to increase activation to bilateral prefrontal cortex. Two sessions per week.
  Interventions: Procedure: Near infrared spectroscopy neurofeedback training

INTERVENTIONS:
Procedure: Near infrared spectroscopy neurofeedback training

SUMMARY:
Background Attention Deficit Hyperactivity Disorder (ADHD) is one of the most frequently diagnosed behavioural disorders in childhood that requires treatment(3-5% of children). It is an important health problem because it impairs social, educational and occupational performance, and increases the risk of other psychiatric disorders including anxiety, depression and substance misuse. There is no cure for ADHD and standard stimulant medication treatment is at best symptomatic. Moreover, stimulants have side effects and parents are often concerned over the long-term effects. A number of non-drug treatments have been developed but these do not target the brain directly. Neurofeedback Training (NTx) is a new, non-drug treatment that targets the brain directly and that can potentially enhance the control of attention in ADHD. NTx could be a valuable alternative and/or adjunct to standard care.

Aims Although NTx has gained popularity in Europe and the US, more rigorous studies are required to support its implementation in the NHS. We therefore propose a pilot study to establish tolerabilty and safety, and to develop treatment protocols and collect data to design a follow-on controlled NTx trial in ADHD.

Methods We plan an open label, single arm, treatment trial of near infrared spectroscopy neurofeedback training of frontal lobe activation in school-aged children with ADHD. 48 participants will be recruited over 1 year and will be offered 20 NTx sessions over 10 weeks. Participants will be recruited from Mental Health Services. Primary outcomes will be safety and tolerability and secondary outcomes will include standard clinical behavioural rating scales and the Test Of the Variables of Attention.

DETAILED DESCRIPTION:
ADHD is one of the most frequently diagnosed conditions in childhood and at least half of patients have symptoms that persist into adulthood. It is important to seek effective treatments for ADHD because children with ADHD often do not reach their full potential and are at increased risk of other psychiatric difficulties in childhood, adolescence and adulthood, including disorders of mood, anxiety, conduct and substance misuse.

Increasingly the available evidence suggest that ADHD may be the result of abnormal levels of certain chemicals and altered brain function. Standard treatment with stimulant medications are aimed at the chemical imbalance and whilst they may help some children, they are of limited benefit in others and of no benefit in more than a quarter of children. Parents are often reluctant to consider medication due to concerns over side effects and the unknown longer term effects of these drugs on their children's developing brains and bodies. Non- drug treatments can provide an alternative and/or adjunct that may overcome some of the concerns about the long-term side effects of drugs. Furthermore, the latest guidelines from the National Institute of Clinical Excellence (NICE, 2008) recommend that medication should only be used as a first-line treatment in severe cases of ADHD. In all other cases it is advised that children receive a group treatment programme and that parents or carers receive parent training and education on ADHD. Whilst these guidelines have been welcomed for promoting alternatives to medication for treating ADHD,concerns have been raised about the feasibility and efficacy of the recommended group interventions for children and individual treatments may be easier to implement and more effective for these children. Therefore, although there are a number of treatments for ADHD, they have limitations in terms of efficacy, tolerability, side effects and practicability. There is therefore a clear rational to investigate new treatments that may be superior in efficacy or valuable as additional or alternative treatments.

Several individual, non-drug interventions for ADHD have emerged over the last thirty years. These include at home parental guidance, classroom based teacher intervention, behavioural therapy, herbal treatment and nutritional supplements. Neurofeedback training appears one of the most promising because the technique directly targets brain functioning in key areas. Neurofeedback training (NTx) uses signals directly from the brain to make subjects aware of brain function. It is an established treatment in epilepsy, migraine and stroke rehabilitation. Abnormal brain function (electrical and blood flow) has been consistently demonstrated in ADHD and may therefore be targeted with neurofeedback. These findings have formed the basis for considering NTx as a potential alternative to medication in the treatment of ADHD.

Compelling evidence from recent controlled studies indicate that NTx that uses electric brain signals (EEG) is a useful treatment in ADHD and that the effects last for at least 6 months. Near infrared spectroscopy neurofeedback (NIRS) neurofeedback training (NIRS NTx) is a newer alternative to EEG NTx. It is easier to administer and may require fewer treatment sessions. NIRS can determine changes in brain activity by measuring changes in the amount of oxygen in the brain. Rather than requiring subjects to alter the pattern of electrical brain activity, NIRSNTx trains subjects to alter blood flow in specific brain areas. Abnormal brain blood flow has been demonstrated in ADHD and typically, these abnormalities include reduced activity of brain areas just behind the forehead.

NIRS NTx is a low cost technique and it can be applied at home, clinic or school. NIRS can safely be applied to the head because the low energy light used for the technique do not cause damage to underlying tissues and is less than 5% of the exposure that occurs in ordinary midday sunlight.

NIRSNTx is performed using a laptop computer, spectroscope, sensor headband and headphones. Typically, patients watch a film on the computer screen whilst wearing the sensor headband and headphones. The headband applies two light sources (red and infrared) and a sensor to the skin overlying the brain area of interest. No special preparation of the skin is necessary. The lights shine through the skin and skull into the brain, where it is absorbed in different quantities depending on the amount of oxygen carried in the blood. Some of the light that is not absorbed is reflected back to the sensor. This signal is analysed in the spectroscope and data are sent to the computer where it is interpreted by software that generates the feedback. Increased blood flow results in positive reinforcement (the film clip advances) and reduced blood flow results in negative reinforcement (the film clip stops and a monotone auditory signal is heard). Subjects learn how to spontaneously increase blood flow to the brain region of interest to enjoy uninterrupted viewing of the film clips. Consequently, NIRS can provide realtime biofeedback to subjects regarding blood flow in specific brain areas.

A typical session of NIRS NTx involves 10 minutes of training at two brain sites. In view of known haemodynamic changes in ADHD and the functional neuroanatomy of attentional control, these sites would be the right and left prefrontal areas. Treatment sessions are offered once or twice weekly for between 15 and 48 sessions. There are no published tolerability data, and available reports come from personal communications with clinicians. The only side effect reported is mild headache that is short lived and self-limiting, immediately after training or on the day following, in around 10% of patients. Clinical observations suggest this predicts a good response to NTx.

Neurofeedback treatment mechanism The human brain has a lifelong capacity to adapt to changes by reorganising itself. This ability is called plasticity and partly works through changes in bloodflow. Examples of plasticity in adults include finding that brain activation leads to brain growth, rewiring of neurons following stroke, larger brain areas dedicated to moving the fingers of musicians, and enlargement of certain brain areas in London cab drivers. NIRSNTx may act in part by enhancing the brain's capacity for plasticity.

In summary, available evidence suggests that NIRS NTx appears safe and capable of targeting specific brain areas that show reduced activity in ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ADHD aged 7 to 17 years
* Patient and legal guardian able to communicate in English
* Patient has been living with parent/guardian for at least six months
* Patient attending school for at least 2 days / week
* ADHD as primary disorder with symptoms present for at least 9 months
* Participants on medication treatment for ADHD must have been on a stable dose for 3 months prior to commencement of the treatment

Exclusion Criteria:

* Significant visual or hearing impairment that would preclude use of NIRS- neurofeedback
* Global learning disability, Autism, psychosis, bipolar disorder, depression, suicidal ideation, or another psychiatric disorder requiring treatment with additional psychotropic medication, current substance dependance or regular use, and severe sleep disorders

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rates | 10 weeks
  The primary outcome measure is the percentage of participants who complete 75% of the 20 training sessions offered.

SECONDARY OUTCOMES:
Adverse effects | 10 weeks
  Occurrence and frequency of training related adverse effects.
Attentional and impulsivity measures | 10 weeks
  Test of Variables of attention (TOVA)
Problem behaviour measure | 10 weeks
  Childhood behavioural checklist (CBCL)
Diagnostic and severity measure | 10 weeks
  Swanson, Nolan and Pelham Questionnaire version IV (SNAPIV)
Psychiatric and social function measure | 10 weeks
  Children's Global Assessment Scale. The CGAS is an adaptation of the Global Assessment Scale (GAS) for young people aged 4-16 years
Treatment response assessment | 10 weeks
  CGI (Clinical Global Impression) is a three-item scale used to assess treatment response in psychiatric patients
Study satisfaction questionnaire | 10 weeks
  Measure of satisfaction of participating.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Dannhauser, PhD, Study Director — North Essex Partnerships University NHS Foundation Trust
Locations (1):
- Aylmer House, Harlow, Essex, United Kingdom